CLINICAL TRIAL: NCT05096325
Title: YpsoPump Occlusion Detection Algorithm: Collection of Real-world Data for In-silico Evaluation of a New Software Algorithm to Refine Occlusion Detection in Subjects With Type 1 Diabetes Using Continuous Subcutaneous Insulin Infusion
Status: Completed | Type: Observational
Sponsor: mylife Diabetes Care AG (Industry)
Collaborators: DCB Research AG (Other)
Responsible Party: Sponsor
Other Study IDs: YPU107
Record Dates: First submitted 2021-10-14; First posted 2021-10-27 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-01

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Continuous subcutaneous insulin infusion; mylife™ YpsoPump®; Occlusion detection algorithm
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study pump: Subjects receive a CE-certified mylife™ YpsoPump® insulin pump system that allows detailed logging of pressure data.
  Interventions: Device: YpsoPump® insulin pump system

INTERVENTIONS:
Device: YpsoPump® insulin pump system — The subjects will receive a CE-certified mylife™ YpsoPump® insulin pump system that allows detailed logging of pressure data. Data will then be analysed in silico comparing the new occlusion detection algorithm with the common occlusion detection algorithm.

SUMMARY:
A common difficulty related to the insulin pumps are occlusions of the insulin infusion set (IIS). This study aims to evaluate the performance of a new software algorithm to detect catheter-occlusion in silico in order to refine the current automated occlusion detection algorithm of the mylife™ YpsoPump®.

ELIGIBILITY:
Inclusion Criteria:

1. Written Informed Consent
2. Subject is diagnosed with T1D
3. Subject on CSII (except patch pumps) for at least 6 months
4. Subject using any type of insulin approved for mylife™ YpsoPump®: Fiasp®, NovoRapid®, Humalog®, Apidra®, Lispro Sanofi
5. Subject using a CGM system for at least 6 months
6. Age ≥ 18
7. Subject willing to continue CSII with mylife™ YpsoPump® during the study
8. Subject willing to use CGM system during the study
9. If the subject wants to use the CGM smartphone app instead of a receiver: Subject ensures to use a compatible smartphone and is willing to share CGM for the duration of the study
10. HbA1c < 9.5% (based on last measurement by treating physician)

Exclusion Criteria:

1. Known allergy/hypersensitivity to medical grade adhesives and/or to physical activity tracker material
2. Known severe nickel allergies
3. History of frequent catheter abscesses associated with pump therapy
4. Treatment with > 1000 mg of acetaminophen every 6 hours
5. Treatment with hydroxyurea
6. Serious acute or chronic disease besides diabetes mellitus or an anamnesis which might, in the opinion of the investigator, pose a risk to the subject, e.g. seizure disorder, adrenal disorder, dialysis for renal failure, cystic fibrosis, active infection
7. Severe late complications of diabetes mellitus, e.g. severe macro- and/or micro-angiopathy (as determined by the investigator)
8. Known hypoglycaemia unawareness
9. Occurrence of self-reported severe hypoglycaemia event requiring third-party assistance within the last 6 months prior to study start
10. Occurrence of self-reported diabetic ketoacidosis requiring healthcare assistance within the last 6 months prior to study start
11. Participation in another investigation with an investigational drug or a pre-market medical device within the 30 days preceding and during the present investigation
12. Female subjects: pregnancy, lactation period, lack of a negative urine pregnancy test (except in case of menopause, sterilization or hysterectomy), or unwilling to use a contraception during the study (for sexually active subjects of childbearing potential)
13. Dependency from the sponsor or the clinical investigator
14. Inability to follow the procedures of the investigation, e.g. due to language problems, psychological disorders, dementia, etc. of the subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target study population consists of adult active users of CSII.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Difference in the number of occlusion alarms generated by the new software algorithm compared to the currently implemented occlusion detection system. | 28 days
  The primary outcome is the difference in the number of occlusion alarms generated by the new software algorithm compared to the currently implemented occlusion detection system throughout the study phase (28 days). The currently implemented method is considered as reference test. Missed alarms using the FIR filter algorithm are considered as false negative alarms while any additional alarm that is detected by the FIR filter algorithm but that was not triggered by the current reference method is considered as false positive.

SECONDARY OUTCOMES:
Retrospective description of the number of occlusions detected including the FIR Filter evaluation | 28 days
  The retrospective description of the number of occlusions detected including the FIR Filter evaluation according to type of insulin, low total daily insulin (≤25U/d) and type of infusion set (micro vs soft) is based on data collected at enrolment and in patients' diaries during follow-up regarding these three characteristics.
Qualitative evaluation of the false positive alarms | 28 days
  The qualitative evaluation of the false positive alarms occurs with the aid of CGM data, movement data collected with a physical activity tracker and the amount of administered insulin over time. The qualitative exploration will be performed by the PIs or delegated members of the study team. They will assess visually and independently each potentially false positive alarm to determine if the alarm qualifies as correct alarm. This qualitative exploration can contribute to future refinements of the occlusion alarm system of the mylife™ YpsoPump®.
Qualitative assessement of the state of the adhesive tapes after study completion | 28 days
  The study subjects will be asked to take pictures of each infusion set prior to change to document the status of the plaster prior to removal. The sponsor will qualitatively assess the state of the adhesive tapes after study completion.

CONTACTS AND LOCATIONS:
Overall Officials: Ingo Braun, Study Director — mylife Diabetes Care AG
Locations (2):
- Institut für Diabetes-Technologie, Forschungs- und Entwicklungsgesellschaft mbH an der Universität Ulm, Ulm, Germany
- Universitätsklinik für Diabetologie, Endokrinologie Ernährungsmedizin & Metabolismus, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No